CLINICAL TRIAL: NCT00756041
Title: An Open-Label, Multi-Center Study to Evaluate the Safety of Long-Term Administration of TAK-128 in Subjects With Mild to Moderate Diabetic Peripheral Neuropathy
Brief Title: Safety Study of TAK-128 in Subjects With Diabetic Peripheral Neuropathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Efficacy.
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-05-TL-128-006; U1111-1128-5801 (Registry Identifier: WHO)
Record Dates: First submitted 2008-09-17; First posted 2008-09-19 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Diabetic Neuropathies
Keywords: Diabetic Mononeuropathy; Diabetic Neuralgia; Mononeuropathy, Diabetic; Neuralgia, Diabetic; Diabetic Polyneuropathy; Drug Therapy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAK-128 100 mg QD (Experimental)
  Interventions: Drug: TAK-128

INTERVENTIONS:
Drug: TAK-128 — TAK-128 100 mg tablet, orally, once daily for up to 1 year.

SUMMARY:
The purpose of this study is to determine the safety of TAK-128, once daily (QD), for treatment of diabetic peripheral neuropathy

DETAILED DESCRIPTION:
Polyneuropathy is a frequent complication of diabetes; it affects most individuals after prolonged hyperglycemia, and diabetic neuropathy is very common in the developed world. Chronic, insidious, distal sensorimotor polyneuropathy with autonomic impairment is the most typical form of diabetic neuropathy. Less common, but more florid presentations include autonomic symptoms or painful neuropathy. Although many patients have no or relatively few symptoms, the chronic polyneuropathy and autonomic dysfunction predispose to neurotrophic foot ulceration; consequently, diabetes is the leading cause of amputation today.

Diabetic neuropathy is a dying-back polyneuropathy with distal degeneration of the longest nerve fibers advancing in a centripetal direction. Multiple histopathological changes are observed, but progressive fiber loss is the hallmark of diabetic polyneuropathy. Other important features include endothelial cell basement membrane thickening, segmental demyelination and remyelination, and axonal atrophy. Similar pathological changes are observed in type 1 and type 2 diabetes. The severity of neuropathy as indicated by the stage of nerve fiber loss determines the clinical, electrophysiological, and quantitative sensory threshold features of this disorder. The functional measures of electrophysiological and quantitative sensory thresholds reflect the morphological changes and the clinical features.

Diabetic polyneuropathy is etiologically related to prolonged hyperglycemia with multiple consequences. Although strict glycemic control prevents neuropathy in type 1 patients if maintained for many years, similar interventions in those with type 2 diabetes mellitus are less successful. Type 2 patients may have neuropathy with considerable nerve fiber loss at the time of diagnosis because of unsuspected hyperglycemia in preceding years. Reversal of established neuropathy with strict glycemic control is not certain to occur, even if maintained for many years. Co-morbid disease often interferes with strict management of type 2 diabetes. Even among those with type 1 diabetes, a minority of patients are successful in maintaining prolonged euglycemia.

TAK-128 is a novel synthetic compound being developed as a treatment for diabetic neuropathy. Subjects participating in this study successfully completed Protocol 01-04-TL-128-003, and earlier study of TAK-128.

ELIGIBILITY:
Inclusion Criteria:

* Has successfully completed protocol 01-04-TL-128-003.
* Female subjects of childbearing potential must be nonpregnant, nonlactating and on an acceptable form of contraception.
* Must be in good health at Enrollment, as determined by a physician at the Month 6 Visit of Protocol 01-04-TL-128-003 (ie, via medical history and physical examination).
* Has clinical laboratory evaluations within the normal reference range for the testing laboratory, unless the results are deemed not clinically significant by the investigator or sponsor, at the Month 6 Visit of Protocol 01-04-TL-128-003.
* Has a creatinine level less than or equal to 2 mg/dL or 176.8 umol/L.
* The subject is willing to follow an American Diabetes Association or similar recommended dietary regimen.

Exclusion Criteria:

* Has developed other neuropathies due to causes other than diabetes such as alcohol abuse liver or renal disease, uremia, toxic exposure, genetic factors, inflammatory demyelinating diseases, monoclonal gammopathies; or endocrine, metabolic or nutritional disorders (included treated or untreated pernicious anemia).
* Has a systolic blood pressure greater than 160 mm HG or diastolic blood pressure is greater than 95 mm HG.
* The subject has an alanine aminotransferase level of greater than 1.5 times the upper limit of normal, active liver disease, or jaundice.
* Has a significant, actively treated or unstable pulmonary, cardiovascular, gastrointestinal, hepatic, hematologic, musculoskeletal, or endocrine (other than diabetes mellitus or stably treated hypothyroidism) disease.
* Cannot use any of the following prescription medications throughout the duration of the study, including:

  * Lipoic acid.
  * Linolenic acid (primrose oil).
  * Inositol.
  * Topiramate.
  * Acetyl-L-Carnitine.
  * Nerve growth factors.
  * Capsaicin.
* Has any other serious disease or condition at the Month 6 Visit of Protocol 01-04-TL-128-003 or at the Baseline/Rollover Visit that might affect life expectancy or make it difficult to successfully manage and follow the subject according to the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2005-09; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent adverse events, vital signs and physical examination findings. | At each visit
Clinical Laboratory Tests (Hematology, Chemistry and Urinalysis). | At each visit
Electrocardiogram results. | At each visit
Weight. | At each visit

SECONDARY OUTCOMES:
Change from Baseline in composite nerve conduction velocities (Electrophysiologic Studies). | Months 6 and 12 or Final Visit
Change from Baseline in the electrophysiologic parameters for individual nerves, including amplitudes (Nerve Conduction Studies). | Months 6 and 12 or Final Visit
Change from Baseline in vibration perception threshold measurements (Quantitative Sensory Testing). | Month 3, 6, 9 and 12 or Final Visit
Change from Baseline in neurological examination (Clinical Neurologic Examination). | Month 3, 6, 9 and 12 or Final Visit
Change from Baseline in pain scores (Short-Form McGill Pain Questionnaire). | Month 3, 6, 9 and 12 or Final Visit
Change from Baseline in quality of life index as assessed by the Short-Form, 36-Item Health Survey. | Month 3, 6, 9 and 12 or Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Medical Director Clinical Science, Study Director — Takeda